CLINICAL TRIAL: NCT00006464
Title: Phase I Dose Escalation Study of UCN-01 (NSC 638850) Plus Cisplatin in Advanced Malignant Solid Tumors
Brief Title: UCN-01 and Cisplatin in Treating Patients With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068274; U01CA062505 (NIH); P30CA033572 (NIH); CHNMC-PHI-28; NCI-T99-0065
Record Dates: First submitted 2000-11-06; First posted 2003-05-30 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — 7-hydroxystaurosporine; Cisplatin

INTERVENTIONS:
Drug: 7-hydroxystaurosporine
Drug: cisplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of UCN-01 and cisplatin in treating patients who have advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of cisplatin when administered with UCN-01 in patients with advanced solid tumors.
* Assess the toxicity and potential antitumor activity of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study of cisplatin.

Patients receive cisplatin IV over 1 hour on day 1 and UCN-01 IV continuously over 36-72 hours beginning on day 2. Treatment continues every 4 weeks for a total of 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 patients receive escalating doses of cisplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 2-3 months for at least 1 year.

PROJECTED ACCRUAL: A total of 9-30 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced or metastatic solid tumor incurable by surgery or other standard therapy
* Tumor site accessible by biopsy
* No brain metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 4,500/mm3
* Absolute neutrophil count at least 2,000/mm3
* Platelet count at least 150,000/mm3

Hepatic:

* Bilirubin normal
* SGOT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine normal
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No New York Heart Association class III or IV congestive heart failure

Other:

* No peripheral neuropathy greater than grade I
* No history of allergic reactions to diuretics or antiemetics (e.g., 5-HT3 antagonists) that would preclude study
* No other uncontrolled illness that would preclude study, including intolerance to vigorous hydration
* No medical, social, or psychological factors that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered
* No greater than 2 prior chemotherapy regimens
* Prior cisplatin allowed if cumulative dose no greater than 400 mg/m2

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Recovered from any prior surgery

Other:

* At least 30 days since prior investigational drugs
* No other concurrent investigational drugs
* No other concurrent anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03; Primary Completion 2005-01 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Gandara, MD, Study Chair — University of California, Davis
Locations (4):
- United States (4):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - City of Hope Medical Group, Pasadena, California
  - University of California Davis Cancer Center, Sacramento, California
  - Norris Cotton Cancer Center, Lebanon, New Hampshire

REFERENCES:
- [Result] Lara PN Jr, Mack PC, Synold T, Frankel P, Longmate J, Gumerlock PH, Doroshow JH, Gandara DR. The cyclin-dependent kinase inhibitor UCN-01 plus cisplatin in advanced solid tumors: a California cancer consortium phase I pharmacokinetic and molecular correlative trial. Clin Cancer Res. 2005 Jun 15;11(12):4444-50. doi: 10.1158/1078-0432.CCR-04-2602. PMID 15958629